CLINICAL TRIAL: NCT01576432
Title: Non-pharmacological Analgesia During Heel Prick: A Randomized, Controlled Trial
Brief Title: Non-pharmacological Analgesia During Heel Prick
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The data showed that pain was higher for our standardized method of sampling
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Miguel Angel Marin Gabriel, Medical Doctor, Pediatrician, Principal Investigator., Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 260 271110
Record Dates: First submitted 2012-04-02; First posted 2012-04-12 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Pain; Breastfeeding
Keywords: Pain; Breastfeeding; Heel prick; Sucrose; Skin-to-skin contact; Newborn
MeSH Terms: conditions — Pain; Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Breastfeeding + skin-to-skin contact (Experimental): In group 1 (BF+SSC), neonates dressed with a diaper were held in prone, in SSC with the mother; breastfeeding (BF) was started at least 5 minutes before heel lance and maintained during sampling
  Interventions: Behavioral: Assess pain with the NIPS score
- Sucrose + skin-to-skin contact (Experimental): In group 2 (sucrose + SSC), neonates were held in prone between the mothers' breast at least 5 minutes before sampling and 2 ml 24% sucrose was given with a sterile syringe in the mouth 2 minutes before heel lance.
  Interventions: Behavioral: Assess pain with the NIPS score
- Skin-to-skin contact (Experimental): In group 3 (SSC), neonates were held between the mother's breast as in group 2, but no sucrose was given.
  Interventions: Behavioral: Assess pain with the NIPS score
- Sucrose (Active Comparator): In group 4 (Sucrose), 2 ml 24% sucrose was administered through a sterile syringe in the mouth 2 minutes before heel lance to neonates laid on supine on a cot; the procedure was done in the presence of the mother
  Interventions: Behavioral: Assess pain with the NIPS score

INTERVENTIONS:
Behavioral: Assess pain with the NIPS score — In group 1 (BF+SSC), neonates dressed with a diaper were held in prone, in SSC with the mother; BF was started at least 5 minutes before heel lance and maintained during sampling. In group 2 (sucrose + SSC), neonates were held in prone between the mothers' breast at least 5 minutes before sampling and 2 ml 24% sucrose was given with a sterile syringe in the mouth 2 minutes before heel lance. In group 3 (SSC), neonates were held between the mother's breast as in group 2, but no sucrose was given. In group 4 (Sucrose), 2 ml 24% sucrose was administered through a sterile syringe in the mouth 2 minutes before heel lance to neonates laid on supine on a cot; the procedure was done in the presence of the mother. Mothers were allowed to speak or touch their babies in all the groups.

SUMMARY:
Objective

To investigate the analgesic effect (measured with NIPS) of breastfeeding in addition to skin-to-skin contact versus other methods of non-pharmacological analgesia during blood sampling through heel lance in healthy term neonates. The influences of non-pharmacological methods on crying time, percentage of crying while sampling, heart rate, number of attempts and duration of sampling were studied.

Methods

Randomised controlled trial performed on 136 healthy term newborns in the maternity ward of a tertiary hospital. The inclusion criteria were: healthy term neonates, wish to breastfeed and absence of feeding during the previous 60 minutes. Neonates were randomly assigned to four groups: group 1, breastfed with skin-to-skin contact ; group 2, oral sucrose with skin-to-skin contact ; group 3, skin-to-skin contact ; or group 4, receiving oral sucrose Data for the primary objective was analysed per intention to treat. This study was approved by local ethical committee.

DETAILED DESCRIPTION:
Healthy term newborns commonly undergo painful procedures even if they do not need intensive care. Heel lance for neonatal screening is the most frequent standardized painful procedure performed in these newborns. Until recently, analgesics were rarely administered to neonates because it was believed that they were less sensitive to pain than more mature infants but current studies suggest that newborns are able to perceive pain. Regardless of the available evidence, appropriate systematic analgesia in common painful procedures in neonates is far from adequate.

Painful stimuli in neonates may have short-term physiologic (increase in intracranial pressure, increase in heart rate or decrease in oxygen saturation) and behavioural consequences (cry, eye squeeze); as well as long-term consequences (altered of pain response in later infancy). Different non-pharmacological methods of analgesia, such as sucrose, skin-to-skin contact (SSC), breastfeeding(BF) or music10, have been used to reduce pain in neonates undergoing venipuncture or heel lancing, and different physiologic pathways to explain the underlying mechanism have been proposed.

A variety of valid and reliable pain assessment instruments have been developed over the past decades. Yet, behavioural pain assessment remains challenging and controversial due to the lack of a gold standard for neonatal pain expression. The Neonatal Infant Pain Scale (NIPS) and the Premature Infant Pain Profile (PIPP) were selected by an international consensus neonatal pain group for acute procedural pain in neonates.

Our main objective was to investigate the analgesic effect (measured with NIPS) of breastfeeding in addition to SSC versus other methods of non-pharmacological analgesia during blood sampling through heel lance in healthy term neonates. Furthermore, the influences of non-pharmacological methods on crying time, percentage of crying while sampling, heart rate, number of attempts and time of sampling were studied.

METHODS

Protocol

This randomised controlled trial was performed on 136 healthy term newborns in the maternity ward of a tertiary hospital. The inclusion criteria were as follows: healthy term neonates (37-416 weeks of gestation) confirmed through a routine physical exam during the first 24h of life, wish to breastfeed and absence of feeding during the previous 60 minutes. Exclusion criteria were as follows: maternal use of opioids, birth in general anesthesia, artificial feeding, previous capillar or venous sampling, and previous admission to the neonatal unit.

Written informed consent was asked to parents during consultation. Study protocol and informed-consent forms were approved by the local ethics committee.

Intervention

Participating neonates were randomly assigned to four groups: group 1, breastfed with SSC (n=35); group 2, receiving oral sucrose with SSC (n=35); group 3, being held in SSC (n=33); or group 4, receiving oral sucrose (n=33). Randomisation was by closed envelopes and nurses and parents were masked to the randomization group but not blinded to the treatment assignment. In group 1 (BF+SSC), neonates dressed with a diaper were held in prone, in SSC with the mother; BF was started at least 5 minutes before heel lance and maintained during sampling. In group 2 (sucrose + SSC), neonates were held in prone between the mothers' breast at least 5 minutes before sampling and 2 ml 24% sucrose was given with a sterile syringe in the mouth 2 minutes before heel lance. In group 3 (SSC), neonates were held between the mother's breast as in group 2, but no sucrose was given. In group 4 (Sucrose), 2 ml 24% sucrose was administered through a sterile syringe in the mouth 2 minutes before heel lance to neonates laid on supine on a cot; the procedure was done in the presence of the mother. Mothers were allowed to speak or touch their babies in all the groups. The standardized procedure of heel prick in our hospital is such as described in group 4.

Throughout the duration of the test, babies were continuously recorded with a video camera at least 2 minutes before sampling and 2 minutes after the procedure. The heel was warmed up by a glove with lukewarm water at least 2 minutes before the sample. Heel lance was made with an automated piercing device for routine neonatal screening for congenital disorders at 48 hours of life. Heart rate was monitored by a pulse oximeter (Radical MasimoSet Datascope, Masimo Corporation, Irvine, CA) set on the infant's hand or foot. Hear rate was measured continuously but special attention was given to three time points: t0 (2 minutes before sampling); t1 (the highest value of the first 10 seconds after heel prick); and t2 (2 minutes after the procedure).

Blood sampling was performed through a standardized procedure by five experienced nurses, who obtained 5 dried spots of blood collected on a filter paper card. If the sample was not enough to complete all of the dried spots on the filter card, a new heel lance was practiced in few seconds. In this case, neonates were assessed for NIPS measure only after the first heel lance; secondary outcomes were evaluated during the whole sampling. Crying time was defined as the duration of crying while sampling. Percentage of crying was defined as the ratio between crying time while sampling and time of the procedure.

Pain scale

The NIPS scale is a validated 6-indicator scale for the assessment of acute pain in neonates11,13. It measure movement of arms and legs, breathing patterns, cry, facial expression and state of arousal. Score ranges from 0 (no pain) to 7 (severe pain). NIPS score <4 means no pain-mild pain. NIPS score ≥4 means moderate-severe pain. NIPS score was measured at three time points: NIPS0 (2 minutes before sampling); NIPS1 (the highest value of the scale in the first 10 seconds after heel prick); and NIPS2 (2 minutes after the procedure). NIPS2 was not recorded if sampling had not finished at this time point. This took place in one newborn (2,8%) of group 1, five (14,2%), six (18.1%), and five (15.1%) of group 2, 3 and 4 respectively. NIPS was measured by three researchers who watched the videos: one expert neonatologist (Observer 1) and two young paediatricians (Observers 2 and 3). Coincidence was 90.8% (95% CI 87.8-93.8) between observers 1 and 2; 75% (70.5-79.5) between observers 1 and 3; and 78.7% (74.7-82.9) between observers 2 and 3. Consequently, only data of the expert neonatologist is shown.

Statistical Analysis

A sample size of 67 infants in each group was calculated to achieve a power of 80% with an α of 0.05 to detect a 0.5-point difference in the NIPS score (assuming SD=1). We decided to make a mid-point analysis when half of the neonates were recruited in order to detect if any of the analgesic methods was better than the standard procedure, and thus modify our clinical practice.

Results were expressed as mean ± standard deviation (SD). Categorical variables were analysed with the χ2 test and the Fisher test. We compared mean between groups with the t-test, ANOVA test and Bonferroni test. We used Mann-Whitney U test, non-parametric ANOVA and Kruskal-Wallis to compare median between groups. The SPSS v.14.0 software package was used to perform all statistical analysis (SPSS Inc. IL, USA). A p-value of 0.05 was considered a statistically significant level of difference. The analysis of the main objective was conducted on an intention-to-treat. Secondary objectives were analysed according to protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term neonates (37-41+6 weeks of gestation) confirmed through a routine physical exam during the first 24h of life
* Wish to breastfeed
* Absence of feeding during the previous 60 minutes.

Exclusion Criteria:

* Maternal use of opioids.
* Birth in general anesthesia.
* Artificial feeding.
* Previous capillar or venous sampling.
* Previous admission to the neonatal unit.

Ages: 37 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
NIPS score during heel prick in healthy term neonates | Midpoint analysis will be conducted when half the patients are recruited (134 subjects), at an estimated time of 12 months.
  The NIPS scale is a validated 6-indicator scale for the assessment of acute pain in neonates. Score ranges from 0 (no pain) to 7 (severe pain).
  NIPS score was evaluated at three time points (2 minutes before heel prick (NIPS-t0), during heel prick (NIPS-t1) and 2 minutes after heel lance (NIPS-t2))in 4 groups where different methods of non-pharmacological analgesia were applied. Results are shown as mean+-SD.
  NIPS score ≥4 means moderate-severe pain. Thus results are also shown as the % of patients with NIPS score ≥4 at different time points (t0, t1 and t2)

SECONDARY OUTCOMES:
Crying time during heel prick in healthy term neonates | Midpoint analysis will be conducted when half the patients are recruited (134 subjects), at an estimated time of 12 months.
  Crying time (in seconds) in 4 groups where different methods of non-pharmacological analgesia were applied. The timer was started at heel prick and stopped when 5 dried spots of blood were collected on a filter paper card. Results are shown as mean+-SD.
Percentage of crying during heel prick in healthy term neonates | Midpoint analysis will be conducted when half the patients are recruited (134 subjects), at an estimated time of 12 months.
  Percentage of crying in 4 groups where different methods of non-pharmacological analgesia were applied during heel prick. Percentage of crying was defined as the ratio between crying time while sampling and time of the procedure. Results are shown as mean+-SD.
Heart rate during heel prick in healthy term neonates | Midpoint analysis will be conducted when half the patients are recruited (134 subjects), at an estimated time of 12 months.
  Heart rate was monitored by a pulse oximeter (Radical MasimoSet Datascope, Masimo Corporation, Irvine, CA) set on the infant's hand or foot. Hear rate was measured continuously but special attention was given to three time points: t0 (2 minutes before sampling); t1 (the highest value of the first 10 seconds after heel prick); and t2 (2 minutes after the procedure). Results are shown as Mean+-SD
Sampling duration during heel prick in healthy term neonates | Midpoint analysis will be conducted when half the patients are recruited (134 subjects), at an estimated time of 12 months.
  Sampling duration (in seconds) was defined as the time spent to obtained 5 dried spots of blood collected on a filter paper card. Results are shown as mean+-SD.
Number of attempts during heel prick | Midpoint analysis will be conducted when half the patients are recruited (134 subjects), at an estimated time of 12 months.
  Number of attempts need to obtaine 5 dried spots of blood collected on a filter paper card. Results are shown as % of patients with 1 attempt and % of patients with 2 attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Marín Gabriel, MD, Principal Investigator — Deparment of Pediatrics. Hospital Universitario Puerta de Hierro-Majadahonda. Madrid. Spain
Locations (1):
- Hospital Universitario Puerta de Hierro-Majadahonda, Madrid, Madrid, Spain

REFERENCES:
- [Background] Porter FL, Wolf CM, Gold J, Lotsoff D, Miller JP. Pain and pain management in newborn infants: a survey of physicians and nurses. Pediatrics. 1997 Oct;100(4):626-32. doi: 10.1542/peds.100.4.626. PMID 9310516
- [Background] Perapoch Lopez J, Pallas Alonso CR, Linde Sillo MA, Moral Pumarega MT, Benito Castro F, Lopez Maestro M, Caserio Carbonero S, de la Cruz Bertolo J. [Developmental centered care. Evaluation of Spanish neonatal units]. An Pediatr (Barc). 2006 Feb;64(2):132-9. doi: 10.1157/13084172. Spanish. PMID 16527065
- [Background] Anand KJ. Clinical importance of pain and stress in preterm neonates. Biol Neonate. 1998;73(1):1-9. doi: 10.1159/000013953. PMID 9458936
- [Background] Mainous RO, Looney S. A pilot study of changes in cerebral blood flow velocity, resistance, and vital signs following a painful stimulus in the premature infant. Adv Neonatal Care. 2007 Apr;7(2):88-104. doi: 10.1097/01.anc.0000267914.96844.ce. PMID 17605449
- [Background] Lindh V, Wiklund U, Hakansson S. Heel lancing in term new-born infants: an evaluation of pain by frequency domain analysis of heart rate variability. Pain. 1999 Mar;80(1-2):143-8. doi: 10.1016/s0304-3959(98)00215-2. PMID 10204726
- [Background] Grunau RE, Holsti L, Peters JW. Long-term consequences of pain in human neonates. Semin Fetal Neonatal Med. 2006 Aug;11(4):268-75. doi: 10.1016/j.siny.2006.02.007. Epub 2006 Apr 24. PMID 16632415
- [Background] Slater R, Cornelissen L, Fabrizi L, Patten D, Yoxen J, Worley A, Boyd S, Meek J, Fitzgerald M. Oral sucrose as an analgesic drug for procedural pain in newborn infants: a randomised controlled trial. Lancet. 2010 Oct 9;376(9748):1225-32. doi: 10.1016/S0140-6736(10)61303-7. PMID 20817247
- [Background] Marin Gabriel MA, Lopez Escobar A, Galan Redondo M, Fernandez Moreno I, del Cerro Garcia R, Llana Martin I, de la Cruz Bertolo J, Lora Pablos D. [Evaluation of pain in a neonatal intensive care unit during endocrine-metabolic tests]. An Pediatr (Barc). 2008 Oct;69(4):316-21. doi: 10.1157/13126555. Spanish. PMID 18928698
- [Background] Bilgen H, Ozek E, Cebeci D, Ors R. Comparison of sucrose, expressed breast milk, and breast-feeding on the neonatal response to heel prick. J Pain. 2001 Oct;2(5):301-5. doi: 10.1054/jpai.2001.23140. PMID 14622809 (Retraction: PMID 14622684 J Pain. 2003 Sep;4(7):415)
- [Background] Hartling L, Shaik MS, Tjosvold L, Leicht R, Liang Y, Kumar M. Music for medical indications in the neonatal period: a systematic review of randomised controlled trials. Arch Dis Child Fetal Neonatal Ed. 2009 Sep;94(5):F349-54. doi: 10.1136/adc.2008.148411. Epub 2009 May 28. PMID 19477913
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Background] Stevens B, Johnston C, Petryshen P, Taddio A. Premature Infant Pain Profile: development and initial validation. Clin J Pain. 1996 Mar;12(1):13-22. doi: 10.1097/00002508-199603000-00004. PMID 8722730
- [Background] Anand KJ; International Evidence-Based Group for Neonatal Pain. Consensus statement for the prevention and management of pain in the newborn. Arch Pediatr Adolesc Med. 2001 Feb;155(2):173-80. doi: 10.1001/archpedi.155.2.173. PMID 11177093
- [Background] Overgaard C, Knudsen A. Pain-relieving effect of sucrose in newborns during heel prick. Biol Neonate. 1999 May;75(5):279-84. doi: 10.1159/000014105. PMID 10095141
- [Background] Leslie A, Marlow N. Non-pharmacological pain relief. Semin Fetal Neonatal Med. 2006 Aug;11(4):246-50. doi: 10.1016/j.siny.2006.02.005. Epub 2006 Apr 24. PMID 16635592
- [Background] Bellieni CV, Bagnoli F, Perrone S, Nenci A, Cordelli DM, Fusi M, Ceccarelli S, Buonocore G. Effect of multisensory stimulation on analgesia in term neonates: a randomized controlled trial. Pediatr Res. 2002 Apr;51(4):460-3. doi: 10.1203/00006450-200204000-00010. PMID 11919330
- [Background] Gibbins S, Stevens B. Mechanisms of sucrose and non-nutritive sucking in procedural pain management in infants. Pain Res Manag. 2001 Spring;6(1):21-8. doi: 10.1155/2001/376819. PMID 11854758
- [Background] Gradin M, Schollin J. The role of endogenous opioids in mediating pain reduction by orally administered glucose among newborns. Pediatrics. 2005 Apr;115(4):1004-7. doi: 10.1542/peds.2004-1189. PMID 15805377
- [Background] Gray L, Miller LW, Philipp BL, Blass EM. Breastfeeding is analgesic in healthy newborns. Pediatrics. 2002 Apr;109(4):590-3. doi: 10.1542/peds.109.4.590. PMID 11927701
- [Background] Codipietro L, Ceccarelli M, Ponzone A. Breastfeeding or oral sucrose solution in term neonates receiving heel lance: a randomized, controlled trial. Pediatrics. 2008 Sep;122(3):e716-21. doi: 10.1542/peds.2008-0221. PMID 18762508
- [Background] Carbajal R, Veerapen S, Couderc S, Jugie M, Ville Y. Analgesic effect of breast feeding in term neonates: randomised controlled trial. BMJ. 2003 Jan 4;326(7379):13. doi: 10.1136/bmj.326.7379.13. PMID 12511452
- [Background] Upadhyay A, Aggarwal R, Narayan S, Joshi M, Paul VK, Deorari AK. Analgesic effect of expressed breast milk in procedural pain in term neonates: a randomized, placebo-controlled, double-blind trial. Acta Paediatr. 2004 Apr;93(4):518-22. doi: 10.1080/08035250410022792. PMID 15188980
- [Background] Castral TC, Warnock F, Leite AM, Haas VJ, Scochi CG. The effects of skin-to-skin contact during acute pain in preterm newborns. Eur J Pain. 2008 May;12(4):464-71. doi: 10.1016/j.ejpain.2007.07.012. Epub 2007 Sep 14. PMID 17869557
- [Background] Johnston CC, Stevens B, Pinelli J, Gibbins S, Filion F, Jack A, Steele S, Boyer K, Veilleux A. Kangaroo care is effective in diminishing pain response in preterm neonates. Arch Pediatr Adolesc Med. 2003 Nov;157(11):1084-8. doi: 10.1001/archpedi.157.11.1084. PMID 14609899
- [Background] Gray L, Watt L, Blass EM. Skin-to-skin contact is analgesic in healthy newborns. Pediatrics. 2000 Jan;105(1):e14. doi: 10.1542/peds.105.1.e14. PMID 10617751
- [Background] Okan F, Ozdil A, Bulbul A, Yapici Z, Nuhoglu A. Analgesic effects of skin-to-skin contact and breastfeeding in procedural pain in healthy term neonates. Ann Trop Paediatr. 2010;30(2):119-28. doi: 10.1179/146532810X12703902516121. PMID 20522298
- [Background] Ludington-Hoe SM, Swinth JY. Developmental aspects of kangaroo care. J Obstet Gynecol Neonatal Nurs. 1996 Oct;25(8):691-703. doi: 10.1111/j.1552-6909.1996.tb01483.x. PMID 8912220
- [Background] Weller A, Feldman R. Emotion regulation and touch in infants: the role of cholecystokinin and opioids. Peptides. 2003 May;24(5):779-88. doi: 10.1016/s0196-9781(03)00118-9. PMID 12895666
- [Background] Weller A, Blass EM. Behavioral evidence for cholecystokinin-opiate interactions in neonatal rats. Am J Physiol. 1988 Dec;255(6 Pt 2):R901-7. doi: 10.1152/ajpregu.1988.255.6.R901. PMID 3202224
- [Background] Blass EM. Behavioral and physiological consequences of suckling in rat and human newborns. Acta Paediatr Suppl. 1994 Jun;397:71-6. doi: 10.1111/j.1651-2227.1994.tb13268.x. PMID 7981477